CLINICAL TRIAL: NCT01918800
Title: A Randomized Trial of a Formal Group Program for Fatigue in Multiple Sclerosis
Brief Title: A Randomized Trial of Two Formal Group Programs for Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: F7777-R
Record Dates: First submitted 2013-08-05; First posted 2013-08-08 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Multiple Sclerosis
Keywords: fatigue; quality of life; rehabilitation; self management; energy effectiveness
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fatigue: Take Control (Experimental): Fatigue: Take Control, is the first formal education program modeled on the MS-related fatigue guideline
  Interventions: Behavioral: Fatigue: Take control
- MS: Take Control (Active Comparator): MS: Take Control includes topics of interest to people with MS other than fatigue.
  Interventions: Behavioral: MS: Take Control

INTERVENTIONS:
Behavioral: Fatigue: Take control — Fatigue: Take Control, is the first formal education program modeled on the MS-related fatigue guideline
  Arms: Fatigue: Take Control
Behavioral: MS: Take Control — MS: Take Control includes topics of interest to people with MS other than fatigue.
  Arms: MS: Take Control

SUMMARY:
The purpose of this study is to compare two different educational programs for people with multiple sclerosis (MS), which is a common and often disabling disease of the central nervous system. MS causes many symptoms including difficulty walking, loss of balance or muscle coordination, fatigue, numbness and tingling and stiffness. The investigators want to determine which program is better at helping improve quality of life and MS symptoms. Both programs use material from the National Multiple Sclerosis Society (NMSS). Both programs include 6 weekly 2-hour class sessions. Up to 600 participants will be enrolled total in 4 VA sites, with about 150 at each site. There will be 10 study visits, all to occur within 11 months. These include 1 baseline visit, 6 two-hour class visits, and 3 follow-up data collection visits. The participants in Portland will also participate in a final 12 month followup visit. Participants will be randomly (by chance) assigned to be part of either group education program. They will have a 1:1 or 50% chance of being in either program.

DETAILED DESCRIPTION:
Treatment of MS-related fatigue represents a significant challenge in providing symptomatic therapy for people with MS. In 1998 the MS Council for Clinical Practice Guidelines published Fatigue and MS, the first evidence based treatment guideline for MS recommending comprehensive treatment for fatigue. This guideline is widely distributed, but does not include a program for implementation. Fatigue: Take Control, is the first formal program modeled on the MS fatigue guidelines. This proposal entails performing a four-center single blind intent-to-treat randomized controlled two-arm parallel design trial of Fatigue: Take Control with MS participants to accomplish three Specific Aims.

Specific Aim #1: Demonstrate that Fatigue: Take Control reduces fatigue in people with MS who are ambulatory and not depressed at the end of the intervention and at three and six months after the intervention compared to a general MS group education program. The primary outcome measure will be the Modified Fatigue Impact Scale (MFIS) chosen for its multi-dimensional nature, recommended use in the Fatigue and MS guideline and sensitivity to change in the pilot study.

Specific Aim #2: Demonstrate that Fatigue: Take Control increases self-efficacy in people with MS who are ambulatory and not severely depressed. Fatigue affects a person's sense of control over his/her life. The investigators will use the MS Self Efficacy Scale (MSSE) for this secondary objective. This measure also demonstrated improvement in the pilot study.

Specific Aim #3: Demonstrate that Fatigue: Take Control results in changes in medication utilization, exercise participation, sleep and health-related quality of life in people with MS who are ambulatory and not depressed. Fatigue affects body functions/structure, activity and participation in all aspects of daily life. Fatigue: Take Control was created with the expectation that fatigue can be reduced by guiding individuals to make the environmental, behavioral and lifestyle changes necessary to manage MS fatigue. This objective will explore important secondary causes of fatigue that impact health-related quality of life by identifying participant changes in: timed walk using the time to walk 25 feet (T25-FW), medication utilization using a self-report medication diary, exercise participation using the self-report Rapid Assessment of Physical Activity (RAPA), sleep quality using the Pittsburgh Sleep Quality Index (PSQI) and changes in overall health-related quality of life using the SF-36.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of MS by 2010 updated McDonald Criteria
* At least 18 years of age
* Able to walk 60 feet without human assistance or architectural support (walls) but with any personal assistive device (cane, crutches, walker) (EDSS-S of 6.5 or less at Visit 1)
* Fluent in written and spoken English, as educational intervention and questionnaires have not been validated in languages other than English.
* Score of greater than 25 on MFIS indicating MS-related fatigue

Exclusion Criteria:

* Severe depression (score on the Beck Depression Inventory II greater than 28)
* Current substance abuse disorder or psychosis
* Any significant uncontrolled medical problem that would limit participation or completion of the study
* MS relapse within the 30 days before screening
* Initiation of new disease modifying treatment within 3 months prior to start of study or participating in an interventional research study
* Current or prior participation in a fatigue management program
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis N Bourdette, MD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (4):
- United States (4):
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Both Portland and Seattle LSIs have opted to send a letter with a copy of the study to participants in the study.

REFERENCES:
- [Result] Hugos CL, Chen Z, Chen Y, Turner AP, Haselkorn J, Chiara T, McCoy S, Bever CT Jr, Cameron MH, Bourdette D; VA MS Fatigue Study Group. A multicenter randomized controlled trial of two group education programs for fatigue in multiple sclerosis: Short- and medium-term benefits. Mult Scler. 2019 Feb;25(2):275-285. doi: 10.1177/1352458517745723. Epub 2017 Dec 11. PMID 29226778
- [Result] Hugos CL, Cameron MH, Chen Z, Chen Y, Bourdette D. A multicenter randomized controlled trial of two group education programs for fatigue in multiple sclerosis: Long-term (12-month) follow-up at one site. Mult Scler. 2019 May;25(6):871-875. doi: 10.1177/1352458518775920. Epub 2018 May 15. PMID 29761722
- [Derived] Knowles LM, Hugos CL, Cameron MH, Haselkorn JK, Bourdette DN, Turner AP. Moderators of Improvements in Fatigue Impact After a Self-management Intervention in Multiple Sclerosis: A Secondary Analysis of a Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Apr 1;101(4):405-409. doi: 10.1097/PHM.0000000000001861. PMID 34347626

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fatigue: Take Control | MS: Take Control
Started | 109 | 109
Completed | 100 | 104
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fatigue: Take Control | MS: Take Control | Total
Number analyzed (Participants) | 109 | 109 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 98 | 96 | 194
  >=65 years | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (9.8) | 53.6 (10.5) | 53.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 77 | 157
  Male | 29 | 32 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 21 | 38
  White | 85 | 80 | 165
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 109 | 109 | 218

OUTCOME MEASURES:

1. Primary Outcome: Modified Fatigue Impact Scale
Description: The self-report, retrospective MFIS measures fatigue symptoms. The full-length MFIS consists of 21 items scored 0-4 for a total score between 0 and 84 and has a coefficient alpha of .81. The MFIS provides a total score and scores for each of three subscales (physical, cognitive and psychosocial) and lower scores on the MFIS and its subscales indicate less fatigue. This is the primary outcome measure for the proposed study and is widely used to assess fatigue in MS.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fatigue: Take Control | MS: Take Control
Number analyzed (Participants) | 109 | 109
units on a scale | 46.1 (12.2) | 46.7 (11.9)
Statistical Analysis 1: Comparison: Fatigue: Take Control vs MS: Take Control; Test type: Superiority or Other; p = .64, paired t test — No adjustment for multiple comparisons. A priori threshold for clinical significance was 7 point improvement

2. Secondary Outcome: Multiple Sclerosis Self Efficacy Scale
Description: The self-report, retrospective MSSE is an 18-item scale of self-efficacy specifically designed for MS patients. This easy to use self-report measure demonstrates internal consistency estimates of about .89 for the full scale and a .75 test-retest correlation. Higher scores on the MSSE indicate higher self-efficacy. Scores range from 180-1800.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fatigue: Take Control | MS: Take Control
Number analyzed (Participants) | 109 | 109
units on a scale | 1434.5 (274.2) | 1352.5 (241.4)
Statistical Analysis 1: Comparison: Fatigue: Take Control vs MS: Take Control; Test type: Superiority or Other; p = 0.04, paired t test — No adjustments for multiple comparisons

3. Secondary Outcome: Beck Depression Inventory II (BDI-II)
Description: The self-report, retrospective BDI-II is a validated 21-item self-report measure of depression widely used in MS studies . Each item is scored between 0 and 3. It is reported to have good reliability (Cronbach's alpha of .81) and validity. Assessing for depression is part of the inclusion/exclusion criteria. Excluding subjects with severe depression is necessary to avoid confounding effects of fatigue and depression. Score range (0-63). Higher scores indicate greater depression.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fatigue: Take Control | MS: Take Control
Number analyzed (Participants) | 109 | 109
units on a scale | 9.5 (7.7) | 10.7 (7.7)
Statistical Analysis 1: Comparison: Fatigue: Take Control vs MS: Take Control; Test type: Superiority or Other; p = 0.35, Paired t test — No adjustment for multiple comparisons

4. Secondary Outcome: SF-36
Description: The SF-36 is a validated measure of health-related quality of life. It is sensitive to change, has appropriate psychometric properties and is frequently used in MS studies. Measures of health-related quality of life are recommended in the systematic review of self-management in neurological disorders. The range for the physical component score is 13.6-61.9. The range for the mental component scores is 15.6-70.0.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fatigue: Take Control | MS: Take Control
Number analyzed (Participants) | 100 | 104
units on a scale
  Physical Composite Score | 24.5 (1.1) | 24.3 (1.1)
  Mental Composite Score | 23.9 (1.7) | 23.8 (1.6)
Statistical Analysis 1: Comparison: Fatigue: Take Control vs MS: Take Control; Test type: Superiority; p = 0.8, Wilcoxon (Mann-Whitney) — The p value in this case is for the SF-36 Physical
Statistical Analysis 2: Comparison: Fatigue: Take Control vs MS: Take Control; The p value in this case refers to the SF-36 Mental; Test type: Superiority; p = .09, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Rapid Assessment of Physical Activity (RAPA)
Description: The self-report, retrospective Rapid Assessment of Physical Activity (RAPA) was developed to provide an easily administered and interpreted means of assessing levels of physical activity among adults older than 50 years. The RAPA is an easy-to-use, valid measure of physical activity for use in clinical practice with older adults. A tool for older adults will be easy to use for people with MS who may not be regular exercisers. Each question has a 'Yes' or 'No' option. The total score of the first seven items is out of 7; participants choose which question corresponds to their activity level. Any score less than 6 is considered suboptimal. From these values we provided a percentage of the number of people exercising optimally in the RAPA Cardiovascular.
  Strength training and flexibility are scored separately (strength training = 1, flexibility = 2, both = 3). Based on total scores we provided a percentage of people at optimum strength and flexibility.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fatigue: Take Control | MS: Take Control
Number analyzed (Participants) | 100 | 104
Participants
  RAPA Cardiovascular | 40 | 33
  RAPA Strength | 51 | 53
  RAPA Flexibility | 69 | 64
Statistical Analysis 1: Comparison: Fatigue: Take Control vs MS: Take Control; Test type: Superiority or Other; p = 0.521, Wilcoxon (Mann-Whitney) — This p value applies to the RAPA Cardiovascular
Statistical Analysis 2: Comparison: Fatigue: Take Control vs MS: Take Control; This p values is for the RAPA Strength; Test type: Superiority; p = 0.4199, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Fatigue: Take Control vs MS: Take Control; Test type: Superiority; p = 0.854, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a l-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score between 0-21. Higher scores indicate worse sleep quality.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fatigue: Take Control | MS: Take Control
Number analyzed (Participants) | 100 | 104
units on a scale | 7.41 (4.27) | 7.71 (3.85)
Statistical Analysis 1: Comparison: Fatigue: Take Control vs MS: Take Control; Test type: Superiority or Other; p = 0.42, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Timed 25 Foot Walk (T25-FW)
Description: The time to walk 8 meters or 25 feet is strongly related to its ordinal counterpart the Ambulation Index (Spearman r = 0.91), without the variability that the ordinal scale reflects.T25-FW was used in this study to measure ambulation status and as an additional measure of mobility. The score for the T25-FWis the average of the two completed trials in seconds
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Fatigue: Take Control | MS: Take Control
Number analyzed (Participants) | 100 | 104
seconds | 8.17 (7.78) | 10.55 (11.94)
Statistical Analysis 1: Comparison: Fatigue: Take Control vs MS: Take Control; Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: Subjects were asked to self report all health problems that occurred during the study at each study visit regardless of relation to study. The study PI then reviewed what subjects had written and categorized each adverse event based on written information from the participant according to organ system class.
Arm/Group | Fatigue: Take Control | MS: Take Control
Serious Adverse Events (participants affected / at risk) | 12/109 | 10/109
Other Adverse Events (participants affected / at risk) | 86/109 | 82/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fatigue: Take Control (N=109) | MS: Take Control (N=109)
MS related (Nervous system disorders) | 1 | 0 — unrelated to research
Surgery (Surgical and medical procedures) | 1 | 0 — unrelated to research
Fracture from a fall (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated to research
Hospitalization for mental health (Social circumstances) | 0 | 1 — unrelated to research
Fracture from a fall (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated to research
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — unrelated to research
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — unrelated to research
Constipation requiring hospitalization (Gastrointestinal disorders) | 1 | 0 — unrelated to research
Defibrulator change resulting in hospitalization (Cardiac disorders) | 0 | 1 — unrelated to research
Bee sting reaction (Immune system disorders) | 1 | 0 — unrelated to research
Hernia (Renal and urinary disorders) | 0 | 1 — unrelated to research
Social circumstances (Social circumstances) | 1 | 0 — unrelated to research
Syncopal event (Nervous system disorders) | 0 | 1 — unrelated to research
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — unrelated to research
Seizure (Nervous system disorders) | 1 | 0 — unrelated to research
MS Hug (Nervous system disorders) | 0 | 1 — unrelated to research
Chest pain (Cardiac disorders) | 0 | 1 — unrelated to research
MS exacerbation (Nervous system disorders) | 1 | 0 — unrelated to research
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Fatigue: Take Control (N=109) | MS: Take Control (N=109)
Chest pain. Undetermined orgin. (Cardiac disorders) | 1 | 0 — unrelated
Shortness of breath and chest pains. (Cardiac disorders) | 0 | 1 — unrelated
nausea-diarrhea (Gastrointestinal disorders) | 1 | 0 — unrelated
Nausea (Gastrointestinal disorders) | 1 | 0 — unrelated
gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 — unrelated
abdominal pain due to gastroparesis (Gastrointestinal disorders) | 0 | 1 — unrelated
bowel discomfort (Gastrointestinal disorders) | 0 | 1 — unrelated
hot flashes (General disorders) | 0 | 1 — unrelated
hot flashes, fatigue and tremors (General disorders) | 0 | 1 — unrelated
vertigo (General disorders) | 0 | 1 — unrelated
Dizziness/balance (General disorders) | 0 | 1 — unrelated
sedation/fainting from side effects of bladder medication (General disorders) | 0 | 1 — unrelated
headache/migraine (General disorders) | 0 | 1 — unrelated
Root canal (General disorders) | 1 | 0 — unrelated
Increase in headaches, vertigo, weakness and fatigue (General disorders) | 0 | 1 — unrelated
Headaches (General disorders) | 0 | 1 — unrelated
headache (General disorders) | 1 | 0 — unrelated
worsening headaches (General disorders) | 1 | 0 — unrelated
sinus infection (Infections and infestations) | 0 | 1 — unrelated
flu (Infections and infestations) | 0 | 1 — unrelated
Infection (Infections and infestations) | 0 | 1 — unrelated
Infection (Infections and infestations) | 1 | 0 — unrelated
fall (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
right hand pain (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
Broken tooth (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
Worsening focus and attention problems (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
Increased pain left side of body (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
fall due to lightheadness (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
pain/stiffness/locking in left hip (from torn ligament) (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
left knee pain (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
right leg weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
increased spasticity (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
swollen foot (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
left arm pain (Musculoskeletal and connective tissue disorders) | 1 | 1 — unrelated
right thigh soreness on ambulation (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
weakenss in right thigh (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
Worsening of left knee. Hyperextension and weakness. (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
strained groin muscle (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
increased shakiness in right arm (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
right hip increased ache, stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
Right arm tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
left shoulder/arm pain into mid back with back spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
Fever, body aches (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
Increase in pain (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
fall (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
Increased pain following car accident (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
heel spur (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 | 0 — unrelated
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 | 1 — unrelated
MS related (Nervous system disorders) | 1 | 0 — unrelated
migraine (Nervous system disorders) | 1 | 0 — unrelated
cluster headaches (Nervous system disorders) | 1 | 0 — unrelated
worsening insomnia (Nervous system disorders) | 1 | 0 — unrelated
MS flareup; 5 days of sterioids (outpatient visits) (Nervous system disorders) | 0 | 1 — unrelated
Insomnia, dizziness, fatigue (Nervous system disorders) | 1 | 0 — unrelated
tremors and increased fatigue (Nervous system disorders) | 1 | 0 — unrelated
changes in peripheral vision (Nervous system disorders) | 1 | 0 — unrelated
chest pain related to MS flare-up (Nervous system disorders) | 0 | 1 — unrelated
fatigue (Nervous system disorders) | 0 | 1 — unrelated
MS exacerbation: leg weakness (Nervous system disorders) | 0 | 1 — unrelated
MS exacerbation: suspected optic neurtits (blurred vision) (Nervous system disorders) | 0 | 1 — unrelated
MS exacerbation:spine curvature, stiffness, spasticity (Nervous system disorders) | 0 | 1 — unrelated
facial numbness (Nervous system disorders) | 0 | 1 — unrelated
Increased leg weakness & declining mobility (Nervous system disorders) | 0 | 1 — unrelated
increased facial pain right side below right eye (Nervous system disorders) | 0 | 1 — unrelated
increased fatigue, spasticity, and tingling. (Nervous system disorders) | 0 | 1 — unrelated
Increased fatigue (Nervous system disorders) | 0 | 1 — unrelated
Left heel drop (Nervous system disorders) | 1 | 0 — unrelated
Mental disorientation (Nervous system disorders) | 1 | 0 — unrelated
epidural steroid injections for pain (Nervous system disorders) | 1 | 0 — unrelated
muscle spasms, neck (Nervous system disorders) | 1 | 0 — unrelated
Diagnosis of external snapping hip syndrome (Nervous system disorders) | 1 | 0 — unrelated
Loss of feeling in vulvar glands (Nervous system disorders) | 1 | 0 — unrelated
Muscle pain (Nervous system disorders) | 1 | 0 — unrelated
excessive fatigue: physical and cognitive change (Nervous system disorders) | 1 | 0 — unrelated
MS related (Nervous system disorders) | 0 | 1 — unrelated
MS related (Nervous system disorders) | 1 | 1 — unrelated
MS related (Nervous system disorders) | 0 | 1/1 — unrelated
UTI (Renal and urinary disorders) | 0 | 1 — unrelated
Recurrent right inguinal hernia (Renal and urinary disorders) | 0 | 1 — unrelated
Angioedema for side effects of bladder medication (Renal and urinary disorders) | 1 | 0 — unrelated
hernia; seen by primary care MD (Renal and urinary disorders) | 1 | 0 — unrelated
bladder issues exacerbated by levoquin antibiotic for bronchitis (Renal and urinary disorders) | 0 | 1 — unrelated
Brusing of uterus, and fallopian tubes (Reproductive system and breast disorders) | 0 | 1 — unrelated
Hemorragic ovarian cysts (Reproductive system and breast disorders) | 0 | 1 — unrelated
vaginal dryness (Reproductive system and breast disorders) | 0 | 1 — unrelated
Breathing/sinus difficutlies from deviated septum surgery (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — unrelated
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — unrelated
sinitus (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — unrelated
Greater difficulty breathing. Cardiac tests negative. Referred to a pulmonologist. (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — unrelated
persistant cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — unrelated
Upper respiratory/cold (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — unrelated
Upper respiratory/cold (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — unrelated
Upper respiratory/cold (Respiratory, thoracic and mediastinal disorders) | 0 | 0 — unrelated
Piece of metal in foot (Skin and subcutaneous tissue disorders) | 1 | 0 — unrelated
skin rash (Skin and subcutaneous tissue disorders) | 1 | 0 — unrelated
Pruritis skin condition (Skin and subcutaneous tissue disorders) | 1 | 0 — unrelated
prutiis skin condition (Skin and subcutaneous tissue disorders) | 0 | 1 — unrelated
skin lesions possible due to injection reaction (Skin and subcutaneous tissue disorders) | 0 | 1 — unrelated
Skin problems (Skin and subcutaneous tissue disorders) | 0 | 1 — unrelated
Skin problems (Skin and subcutaneous tissue disorders) | 1 | 0 — unrelated
Skin problems (Skin and subcutaneous tissue disorders) | 0 | 0 — unrelated
increase in anxiety (Social circumstances) | 0 | 1 — unrelated
Emotional (Social circumstances) | 1 | 0 — unrelated
Emotional (Social circumstances) | 0 | 1 — unrelated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes